CLINICAL TRIAL: NCT05691738
Title: The Effect of Modified Otago Exercises on Metabolic Parameters, Joint Position Sense, Balance and Health-Related Physical Fitness Parameters in Individuals With Diabetic Neuropathy
Brief Title: Effects of Modified Otago Exercises in Individuals With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ali CEYLAN, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU-ACEYLAN-001
Record Dates: First submitted 2022-12-23; First posted 2023-01-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Neuropathy
Keywords: Otago Exercise; Joint Position Sense; Balance; Physical Fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The physician who will evaluate the metabolic parametres will not know which arm the individual is in. İn addition, the participants will not know which arm they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Experimental): Information will be given about diabetes and its complications.Modified Otago Exercise will be applied by the physiotherapist.Participants will be given a home program
  Interventions: Other: Exercise Group
- Control Group (Other): Information will be given about diabetes and its complications.Participants will be given a home program
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Exercise Group — The exercise group will be informed about diabetes and diabetes complications. A total of 16 sessions of 8 weeks, modified otago exercises will be applied individually by the research physiotherapist.Individuals will be allowed to walk at a moderate pace for at least 30 minutes 5 days a week (home program).
  Arms: Exercise Group
Other: Control Group — The control group will be informed about diabetes and diabetes complications. Individuals will be allowed to walk at a moderate pace for at least 30 minutes 5 days a week (home program)
  Arms: Control Group

SUMMARY:
The aim of the study is to investigate the effects of modified otago exercises on joint position sense, balance and physical fitness parameters in individuals with diabetic neuropathy. In addition aim of to examine the effects of exercise on metabolic variables and to gain exercise awareness in diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Neuropathy Diagnosed with Type 2 Diabetes between the Ages of 40-65 Years
* Cooperative, able to take instructions (Mini Mental Test score of 24 and above)
* Able to walk independently
* With a Body Mass Index Below 40 Kg/M2
* Not Doing Regular Physical Activity for the Last 6 Months
* Voluntarily participated in the research

Exclusion Criteria:

* Additional neurological problem other than neuropathy
* Any orthopedic or systemic problems that will prevent him from performing the exercises
* The presence of pathology related to the lower limb that occurred within the last 6 months (surgery, fracture, soft tissue injuries, etc.)
* Pregnant
* Vision problem that cannot be corrected with glasses or lenses
* Hearing loss that cannot be corrected with hearing aids
* Foot ulcer
* Patients who have been diagnosed with cancer and are receiving chemotherapy in this context
* With limitation of the range of motion of the joints of the lower extremities

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Level | Change from baseline at 8 weeks
  Routinely, the glycated hemoglobin (Hba1c) (mg/dL) level will be recorded in the blood laboratory results by the endocrinologist.
Blood Cholesterol Level | Change from baseline at 8 weeks
  Routinely, the cholesterol (mg/dL) level will be recorded in the blood laboratory results by the endocrinologist.
Blood Triglycerides Level | Change from baseline at 8 weeks
  Routinely, the triglycerides (mg/dL) level will be recorded in the blood laboratory results by the endocrinologist.
Blood HDL Cholesterol Level | Change from baseline at 8 weeks
  Routinely, the HDL cholesterol (mg/dL) level will be recorded in the blood laboratory results by the endocrinologist.
Blood LDL Cholesterol Level | Change from baseline at 8 weeks
  Routinely, the LDL cholesterol (mg/dL) level will be recorded in the blood laboratory results by the endocrinologist.
Joint Position Sense Evaluation | Change from baseline at 8 weeks
  Ankle joint position sense of 10 degrees dorsiflexion and 15 degrees plantar flexion target angles will be evaluated.
The Timed Up & Go (Functional Mobility Assessment) | Change from baseline at 8 weeks
  Patients sitting in a chair without armrests will be asked to stand up with the start command and walk the 3-meter distance, whose start and end points are specified before, turn around and sit on the chair again. The test will be repeated 3 times and the average time will be recorded.
Balance Evaluation | Change from baseline at 8 weeks
  Balance Error Scoring System:Practices are performed on hard and soft ground separately in 3 positions, two feet, one foot and tandem stance, with eyes closed.After the test position is taught to the patient, the patient is asked to close their eyes and hold the position for 20 seconds.A mistake made for 20 seconds on each floor and position is recorded as 1 point.The maximum error score is 10.All assessments are made without shoes
Body Mass İndex Evaluation | Change from baseline at 8 weeks
  Body weight of the individual is recorded in kilograms and height in meters.Calculated by dividing body weight by the square of the height in meters (kg/m2)
Body Weight | Change from baseline at 8 weeks
  Calculated in kilograms (kg) with a Tanita BC730 brand scale
Body Fat Percentage | Change from baseline at 8 weeks
  Body fat percentage is calculated as percentage (%) with Tanita BC730 brand scale
Lean Body Weight | Change from baseline at 8 weeks
  Calculated in kilograms (kg) by subtracting body fat from body weight.
Cardio-respiratory Fitness Evaluation | Change from baseline at 8 weeks
  A distance of 30 meters is created in an area measuring 10x40 meters, the start and end points are marked.Patients are asked to walk on the designated line for 6 minutes at the highest speed they can walk without running.At the end of 6 minutes, the distance they have walked is recorded in meters.
Sit and Reach Test (Flexibility ) Evaluation | Change from baseline at 8 weeks
  The patient is asked to lie down without bending his knees towards the ruler placed on the flexibility table. Before the test, the patient is asked to reach forward 1-2 times and is taught what to do. Then the patient is asked to lie forward 3 times and the average of the data obtained is recorded in centimeters.
Muscle Strength (30-second Chair Stand Test) Evaluation | Change from baseline at 8 weeks
  Sitting in a standard chair without armrests, the patient is asked to cross his hands over his shoulder. With the start command, the stopwatch is kept and the patient is asked to stand up completely from the chair and sit down again. The number of repetitive movements for 30 seconds is recorded.
Falling Risk | Change from baseline at 8 weeks
  Fall Efficacy Scale International: It is a common test battery with 16 items that reveals the possibility of falling in patients.The higher the test score, the higher the probability of falling in the patient.

SECONDARY OUTCOMES:
Cognitive Status | a day before the start of treatment
  Mini Mental Test will be used to evaluate the cognitive status of individuals. It is a short, useful, standardized test that provides the opportunity to evaluate cognitive performance in a short time. A high score indicates a good cognitive status. The maximum possible score is 30. A score of 17 and below is considered severe dementia, a score of 18-23 is considered mild dementia, and a score of 24-30 is considered normal.
Neuropathic Pain Scale | Change from baseline at 8 weeks
  Self-Leeds Assesment of Neuropathic Symptoms & Signs Pain Score: It is a simple test used in the differential diagnosis of neuropathic pain at the bedside.A score of 12 and above is diagnostic for neuropathic pain
Individual Exercise İntensity | a day before the start of treatment
  Borg Scale: It is a method used to determine the exercise tolerance of the individual.The individual scores the fatigue she feels between 6-20.Fatigue level; nothing (6), very very light (7-8), very light (9-10), light (11-12), somewhat difficult (13-14), difficult (15-16), very difficult (17- 18), very very difficult (19), exhaustion (20)
Monofilament Evaluation | a day before the start of treatment
  The monofilament is touched to the relevant point on the foot until it takes a C shape. Absence of a 4.17 or thicker monofilament is interpreted as being compatible with neuropathy.Failure to detect a 5.07 monofilament is considered as a loss of protective sensation.
Diaposan (Vibration) Evaluation | a day before the start of treatment
  A 128 Hz tuning fork, which was oscillated before, is placed on the metatarsophalangeal joint of both feet of the individual and the patient is asked to feel the vibration. If the investigator still perceives the vibration as soon as the patient says he does not feel the vibration, it is considered neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: ALİ CEYLAN, MSc, Principal Investigator — Karamanoğlu Mehmetbey University; Ertuğrul DEMİRDEL, PhD, Study Chair — Ankara Yildirim Beyazıt University
Locations (1):
- Karaman Provincial Health Directorate Karaman Training and Research Hospital, Karaman, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No